CLINICAL TRIAL: NCT06626750
Title: Evaluating Stress Management Strategies Within the School Readiness Parenting Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Paulo A. Graziano, PhD, Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-23-0039
Record Dates: First submitted 2024-08-28; First posted 2024-10-04 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Parenting; Stress; Disruptive Behavior Disorder; Parent-Child Relations; ADHD
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional School Readiness Parenting Program (Active Comparator): Parents will be required to attend a School Readiness Parenting Program for 1.5 to 2 hours weekly. Sessions include behavioral management strategies and school readiness. Behavior management strategies are delivered to the entire group via a Community Parent Education Program (COPE) style modeling problem solving approach; parents contribute to the didactic discussion. The behavioral management content is derived from Parent-Child Interaction Therapy (PCIT).
  Interventions: Behavioral: Summer Treatment Program for Pre-Kindergarteners and Kindergarteners; Behavioral: School Readiness Parenting Program (SRPP)
- School Readiness Parenting Program + Cognitive Behavioral Therapy (Experimental): For those randomly assigned to the additional parenting stress modules, parents will receive the same SRPP as well as three additional modules to target parenting stress. The modules will incorporate practices based on Cognitive-Behavioral Therapy (CBT).
  Interventions: Behavioral: Summer Treatment Program for Pre-Kindergarteners and Kindergarteners; Behavioral: School Readiness Parenting Program (SRPP); Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Summer Treatment Program for Pre-Kindergarteners and Kindergarteners — Children will be concurrently enrolled in our Summer Treatment Program for Pre-Kindergarteners and Kindergarteners (STP-PreK/K). The STP-PreK/K simulates a school-like schedule and runs for 7-weeks and last 7 hours/day, Monday through Friday, with periods of seatwork, large/small group activities, circle time, and classroom meetings along with a recreational period. Academic curriculum are individualized depending upon child's current level. The behavioral modification program uses a visual response cost system in which children lose points for not following classroom rules (these rules are operationalized and determined during the development phase). Dots earned are then used for daily and weekly rewards. In addition to the academic and behavioral modification program, one group of children will participate in social-emotional/self-regulation training exercises on a daily basis designed to teach them social skills and how to control their emotions, behaviors, and attention.
Behavioral: School Readiness Parenting Program (SRPP) — The School Readiness Parenting Program (SRPP) helps parents of young children develop skills that support their child's readiness for kindergarten and first grade. It focuses on positive parenting practices that enhance social, emotional, and cognitive development. The sessions cover managing child behaviors, promoting early literacy, and fostering problem-solving skills. Parents learn effective communication, consistent routines, and how to create a supportive home environment.
Behavioral: Cognitive Behavioral Therapy (CBT) — Cognitive Behavioral Therapy (CBT) is a structured, goal-oriented therapy that helps individuals identify and change negative thought patterns and behaviors. It focuses on the link between thoughts, emotions, and actions to improve mental health. Specific to the current project, CBT can reduce stress by teaching parents to reframe unhelpful thoughts, manage challenging emotions, and develop effective coping strategies for difficult situations, leading to more positive parenting experiences.
  Arms: School Readiness Parenting Program + Cognitive Behavioral Therapy

SUMMARY:
The goal of this randomized study is to learn if adding three additional parent training sessions (focused on alleviating parental stress) to an already well-established treatment (School Readiness Parenting Program [SRPP]) in improving outcomes up to 6- and 12-months later for families of children with disruptive behavior disorders. The main questions it aims to answer are:

The primary objective of this protocol is to evaluate the effects of three additional cognitive behavioral therapy (CBT) based parent training sessions to the SRPP to reduce parent stress and improve parent-child interactions.

The secondary objective of this protocol is to evaluate the behavioral, emotional, and physical health-based functioning among young children with ADHD.

Researchers will compare families who receive the SRPP alone to families who receive the SRPP + the three additional CBT focused sessions.

Parents will be sent surveys to complete prior to the baseline assessment via REDCap (online). Parent and child participants will undergo 2 hours of baseline assessments evaluating behavioral, cognitive, and academic functioning as well as parent-child interactions. Parents will provide contact information for their child's teacher and the teacher will sent three surveys to complete online via REDCap.

DETAILED DESCRIPTION:
A total of 120 families will all receive a 7-week behavioral treatment (Summer Treatment Program) for children going into kindergarten or first grade with a disruptive behavior disorder. They will also be randomized to receive either a well-established school readiness parenting program (8 sessions) alone or the same parent training program with three additional parent training sessions (11 sessions). The three additional parent training sessions will include information on parental stress tolerance and cognitive-behavioral skills to improve parent's self-efficacy and sense of competence that are not included in the original school readiness parenting program. Parents will complete questionnaires and lab tasks with their child at baseline, 6-month follow up, and 12-month follow up. Lab tasks include a 15-minute parent-child play-like situation, and a 10-minute "difficult puzzle" task. The results of this research study may improve our understanding of child behavior and early school success and have important implications on parenting programs.

ELIGIBILITY:
Inclusion Criteria:

* At-risk clinical range on the BASC-Preschool Version (per parent and teacher report) or clinical diagnosis of Attention-Deficit/Hyperactivity Disorder and/or Oppositional Defiant Disorder based on the Disruptive Behavior Disorders Scale or the Diagnostic Interview Schedule for Children
* Parent and teacher report of significant levels of impairment at home and at school on the Impairment Rating Scale

Exclusion Criteria:

* Significant sensory impairments (e.g. deafness, blindness)
* Significant motor difficulties that impair mobility (e.g., cerebral palsy)
* Families with current Department of Children and Family (DCYF) involvement

Any family meeting exclusionary criteria will be referred to appropriate intervention services in Miami-Dade County. Children will not be excluded on the basis of race/ethnicity, sex, or socioeconomic status.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Parent Stress Index (PSI) | Baseline, between 4 to 6 months after baseline (post treatment), and 12-months
  A 36-item self-report instrument for parents of children ages 1 month to 12 years containing three subscales (Parent Distress, Parent-Child Dysfunctional Interaction, Difficult Child). Total scores range between 36 to 180, with higher scores indicating higher levels of perceived parenting stress.
Dyadic Parent-Child Interaction Coding System | Baseline, between 4 to 6 months after baseline (post treatment), and 12-months
  A Behavioral coding system that measures the quality of parent-child interactions during three 5-minutes standard situations that vary in the degree of parental control (i.e., parent reading to child, child-led play, parent-led play, and clean-up). Parent verbalizations are coded for positive and negative communication patterns and are totaled at the end of each 5-minute situation.
Difficult Puzzle Lab Task - Early Parenting Coding System (EPCS) | Baseline, between 4 to 6 months after baseline (post treatment), and 12-months
  Co-operative goal-directed interactions between mothers and children will be coded from a video of mother-child interactions in a laboratory task intended to be moderately stressful for the dyad. The EPCS captures a range of parenting behaviors that are typically exhibited in interactions with young children. This coding system consists of nine global ratings. Behaviors are rated on a Likert scale, with scores ranging from low to high (i.e.,1 to 7), with higher scores indicating more positive parenting behaviors.
Cognitive Behavioral Therapy Parent Quiz | Baseline, between 4 to 6 months after baseline (post treatment), and 12-months
  Parents will complete a 25-item multiple choice quiz on cognitive behavioral therapy skills. Scores range from 0% to 100%, with higher percentages indicating greater knowledge of session material.

SECONDARY OUTCOMES:
Behavior Assessment System for Children | Baseline, post treatment, 12-months
  A widely used behavior checklist that taps emotional and behavioral domains of children's functioning. There are three parent versions: Preschool Form (ages 2-5, 134 total items), Child Form (ages 6-11, 160 total items), and Adolescent form (ages 12-21, 150 total items).
Disruptive Behavior Disorders Rating Scale | Baseline, post treatment, 12-months
  Assesses for the presence of Attention-Deficit/Hyperactivity Disorder, Oppositional Defiant Disorder, or Conduct Disorder symptoms . On the DBD, parents are asked to provide ratings of (0) not at all, (1) just a little, (2) pretty much, or (3) very much for each symptom listed.
Treatment Satisfaction Survey | Post treatment
  Parents will complete a 40-item treatment satisfaction survey assessing their child's response to treatment, their attitudes towards the treatment format, and other related outcomes.
SRPP activities practice | During/Post-treatment
  Percentage of weekly activities completed as part of SRPP sessions
Difficult Puzzle Lab Task - Early Parenting Coding System (EPCS) | Baseline, post treatment, 12-months
  Children's emotion dysregulation will be coded during the task via global codes that have been previously used in prior temperament studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified summary data from the study will be shared with other researchers upon request and after completion of study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon completion of study and for 3 years.